CLINICAL TRIAL: NCT00307346
Title: Physiology of Weakness With Movement Disorders
Brief Title: Physiology of Weakness in Movement Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060125; 06-N-0125
Record Dates: First submitted 2006-03-24; First posted 2006-03-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-01-25

CONDITIONS: Movement Disorders
Keywords: Movement-Related Potential; Electroencephalogram; Psychogenic Movement Disorders; Psychogenic Movement Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Movement Disorders

SUMMARY:
This study will compare electroencephalograph (EEG) recordings in healthy volunteers and in people with movement disorders to examine brain activity associated with the weakness. EEG records the electrical activity of the brain ("brain waves").

Healthy volunteers and patients with arm or leg weakness who are between 18 and 80 years of age may be eligible for this study. Healthy subjects are screened with a medical history, physical and neurological examinations, and a questionnaire. They must be right-handed and never have had a neurological disease or head trauma.

All participants have an EEG. An elastic cap with electrodes is placed on the subject's scalp to record the brain's electrical activity. During the EEG, subjects are required to resist against a force with their arm, elbow, shoulder or leg for as long as they can. Several recordings are done with short breaks between them.

DETAILED DESCRIPTION:
Objective

Give way weakness is a symptom often associated with psychogenic etiology, but its neurophysiological basis is poorly understood. Our objective in this study is to identify the cerebral mechanism of give way weakness.

Study population

We will study 6 patients with give way weakness and 6 healthy volunteers all age 18 years old or older.

Design

In this study, patients will try to resist against the examiner's force and subsequently give way. Electroencephalography (EEG) will be recorded while this maneuver is performed repeatedly.

Outcome measures

Movement-related cortical potential (MRCP) analysis will be performed on the data and its amplitude (in volts) and latency (in seconds) in each individual patient will be described in contrast to the data obtained from healthy volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Both patients and healthy volunteers will be between age 18 and 80.
* Patients will be evaluated in the Human Motor Control Clinic at NINDS.
* The definite diagnosis of the disease may not be completely established at the time of recording.
* Patients have clear and reproducible symptoms of give way weakness of either upper or lower extremities.
* Patients have to be able to resist against the examiner for at least two seconds before giving way.
* Healthy volunteers are right handed adults without history of neurological disease or severe head trauma.

EXCLUSION CRITERIA:

* Subjects (patients or volunteers) who cannot understand the instructions and consent forms of the protocol will be excluded.
* Subjects who cannot follow the instruction during the entire recording for whatever reason will be excluded.
* Patients with a documented organic central nervous system lesion may be excluded from the study. This will be discussed in detail for each individual subject at the Human Motor Control Clinic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03-23; Study Completion 2011-01-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Terada K, Ikeda A, Nagamine T, Shibasaki H. Movement-related cortical potentials associated with voluntary muscle relaxation. Electroencephalogr Clin Neurophysiol. 1995 Nov;95(5):335-45. doi: 10.1016/0013-4694(95)00098-j. PMID 7489662
- [Background] Terada K, Ikeda A, Yazawa S, Nagamine T, Shibasaki H. Movement-related cortical potentials associated with voluntary relaxation of foot muscles. Clin Neurophysiol. 1999 Mar;110(3):397-403. doi: 10.1016/s1388-2457(98)00017-0. PMID 10363761
- [Background] Toma K, Honda M, Hanakawa T, Okada T, Fukuyama H, Ikeda A, Nishizawa S, Konishi J, Shibasaki H. Activities of the primary and supplementary motor areas increase in preparation and execution of voluntary muscle relaxation: an event-related fMRI study. J Neurosci. 1999 May 1;19(9):3527-34. doi: 10.1523/JNEUROSCI.19-09-03527.1999. PMID 10212312